CLINICAL TRIAL: NCT02161354
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study To Determine The Efficacy and Safety of Buprenorphine (as NTC-510 and NTC-510A) in Subjects With Pain Following Surgical Extraction of 1 or 2 Third Molars.
Brief Title: Safety and Efficacy Study of NTC-510 to Treat Pain Following Dental Surgery of Third Molars
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: safety and efficacy after cohort 5 did not warrant further dose escalation
Sponsor: NanoSHIFT LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTC-510-004
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Dental Pain
Keywords: Dental Pain; Acute Pain; Mild Pain; Moderate Pain
MeSH Terms: conditions — Toothache; Acute Pain | interventions — Buprenorphine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 2mg dose of NTC-510 or placebo (Experimental): Subjects will be dosed with 2 mg of NTC-510 or placebo.
  Interventions: Drug: NTC-510 capsules; Drug: Placebo Capsules
- 4 mg dose of NTC-510 or placebo (Experimental): Subjects will be dosed as a split dose of 2 mg followed by 2 mg an hour later of NTC-510 or placebo.
  Interventions: Drug: NTC-510 capsules; Drug: Placebo Capsules
- 6 mg dose of NTC-510 or placebo (Experimental): Subjects will be dosed with 6 mg of NTC-510 or placebo.
  Interventions: Drug: NTC-510 capsules; Drug: Placebo Capsules
- 2 mg dose of NTC-510, NTC-510A or placebo (Experimental): Subjects will be dosed with 2mg of NTC-510A or placebo
  Interventions: Drug: NTC-510 capsules; Drug: Placebo Capsules; Drug: NTC-510A Capsules
- 4 mg dose of NTC-510, NTC-510A or placebo (Experimental): Subjects will be dosed with 4 mg of NTC-510A or placebo
  Interventions: Drug: NTC-510 capsules; Drug: Placebo Capsules; Drug: NTC-510A Capsules
- 6 mg dose of NTC-510, NTC-510A or placebo (Experimental): Subjects will be dosed with 6 mg of NTC-510A or placebo
  Interventions: Drug: NTC-510 capsules; Drug: Placebo Capsules; Drug: NTC-510A Capsules

INTERVENTIONS:
Drug: NTC-510 capsules — Subjects will be randomized to one of 3 groups and NTC-510 will be given as a single oral dose of 2.0 mg, a split dose of 2.0 mg followed by 2.0 mg an hour later, or 6.0 mg for acute pain relief (PR) following third molar extraction.
  Other Names: buprenorphine and naloxone capsules
Drug: Placebo Capsules — Subjects will be randomized to one of 3 groups and placebo capsules will be given as a single oral dose of for acute dental pain following third molar extraction.
  Other Names: placebo capsule
Drug: NTC-510A Capsules — Subjects will be randomized to one of 3 groups where NTC-510A or placebo will be given as a single oral dose of 2.0, 4.0, or 6 mg for acute pain relief (PR) following third molar extraction
  Other Names: buprenorphine capsules
  Arms: 2 mg dose of NTC-510, NTC-510A or placebo; 4 mg dose of NTC-510, NTC-510A or placebo; 6 mg dose of NTC-510, NTC-510A or placebo

SUMMARY:
To evaluate the efficacy of a single dose NTC-510 or NTC-510A for dental pain following third molar extraction.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the efficacy, concentration versus efficacy relationship, and safety of NTC-510 and NTC-510A at doses of 2.0, 1.0, and 0.5 mg.

The study will consist of 4 phases: screening (within 28 days before check-in), check-in (before surgery on Day 1), treatment (surgery, randomization, and treatment with study drug on Day 1), and follow up (Days 6 to 8). During the screening phase, screening procedures will be performed, subject eligibility will be determined, and written consent will be obtained. Subjects will then undergo dental surgery to extract 1 or 2 third molars (with at least 1 partial or complete bony mandibular extraction). The impaction score ([1] erupted in tissue, [2] broken soft tissue, [3] partial bony impaction, and [4] full bony impaction) will be collected for statistical adjustment should there be randomization imbalance. The surgery will be conducted according to standard clinical unit procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, understand, and sign the approved informed consent form.
* Subject is an adult between 18 and 45 years of age, inclusive, who has been evaluated and scheduled for an elective third molar surgical extraction (targeting 1 or 2 third molars, at least 1 of which is mandibular and fully or partially impacted by bone). Supernumerary or affected adjacent teeth may be removed at the surgeon's discretion.
* Subject has body mass index of 18.0 to 30.0 kg/m2, inclusive.
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device (copper/hormonal), NuvaRing®, Depo-Provera®, or double-barrier method, and have a negative pregnancy test prior to surgery. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or have had a hysterectomy and/or bilateral oophorectomy.
* Subject must experience moderate to severe pain (i.e., rating of 2 or 3 on a 4-point categorical PI scale [0 = none, 1 = mild, 2 = moderate, and 3 = severe] and a score of ≥ 50 mm on a 100 mm VAS) within 5 hours after the dental extraction.
* Subject has been administered only 2% topical benzocaine, lidocaine with epinephrine, and/or nitrous oxide as preoperative medication.
* Subject is determined by the investigator to be otherwise in good health and unlikely to be at risk from participation in this study.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Subject has a history of human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Subject has participated in any clinical research study within the previous 8 weeks.
* Subject has a history of seizures and/or significant head trauma.
* Subject has an abnormal cardiac condition including any of the following:

  * Medically significant disorders of cardiac rate and/or rhythm
  * QTc interval > 450 msec (calculated using Fridericia's correction) or uncorrected QT interval > 500 msec, PR interval > 240 msec or ≤ 110 msec, evidence of second or third degree atrioventricular block, pathological Q-waves (defined as Q-wave > 40 msec or depth > 0.5 mV), evidence of ventricular pre-excitation, complete left bundle branch block, and/or resting heart rate outside the range of 40 to 120 beats per minute
* Subject has evidence of clinically significant abnormal laboratory values including the following:

  * Impaired kidney function (i.e., serum creatinine ≥ 1.5 mg/dL)
  * Impaired liver function (laboratory test values ≥ 3 times the upper limit of normal [ULN] for aspartate aminotransferase or alanine aminotransferase, or values > 2 times the ULN for alkaline phosphatase), or total bilirubin level > 1.5 times the ULN or, in the opinion of the investigator, liver function impairment to the extent that the subject should not participate in this study
  * Presence of Gilbert's Syndrome or any known hepatobiliary abnormalities
  * Any other laboratory values judged as clinically significant by the investigator
* Subject has a history of chronic or sustained intake of opioid drugs in the preceding 12 months, or has taken any medication containing opioid compounds in the month preceding entry to this trial.
* Subject has a history of alcohol or substance abuse or addiction within 2 years before screening and/or routine consumption of 3 or more alcohol-containing beverages per day. Subject has consumed alcohol within 3 days before administration of study drug or cannot abstain for the duration of confinement to the clinical unit.
* Subject has a prior history of intolerance to opioid drugs, their excipients, or related compounds.
* Subject has positive urine test for alcohol, cotinine, or drugs of abuse at screening or check-in. If a subject is excluded for a positive drug screen due to prescribed medication for pain from an infected molar, the subject may be rescreened after the appropriate washout period.
* Subject has used any medication (with the exception of vitamins and contraceptives), including over-the-counter medications, herbal and/or mineral supplements, dietary supplements, or has ingested grapefruit-containing foods or beverages within 3 days before administration of study drug, or cannot abstain for the duration of confinement to the clinical unit.
* Subject has ingested caffeine-containing foods or beverages (e.g., coffee, tea, chocolate, and colas) within 24 hours before administration of study drug or cannot abstain for the duration of confinement to the clinical unit.
* Subject has smoked or used other nicotine products within 3 days before study drug administration or cannot abstain for the duration of confinement to the clinical unit.
* Subject has the presence of any conditions possibly affecting drug absorption (e.g., gastrectomy or malabsorption) or has taken oral medications that affect gastric acid availability (including H2 antagonists, proton-pump inhibitors, and antacids) within 3 days before administration of study drug.
* Subject has any current dental or medical condition that could prevent safe participation in this study.
* Subject has significant medical or psychiatric symptoms, cognitive impairment, or other factors which, in the opinion of the investigator, would preclude compliance with the protocol, adequate cooperation in the study, or obtaining informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Decrease in dental pain when taking a single doses of NTC-510 or NTC-510A at 2.0, 1.0, or 0.5 mg following third molar extraction. | 24 hours

SECONDARY OUTCOMES:
Evaluate the number of subjects with adverse events following a single oral dose of 2.0, 1.0, or 0.5 mg for acute pain relief (PR) following third molar extraction | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: William L Buchanan, MD,DDS, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Dental Pain Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided